CLINICAL TRIAL: NCT05103306
Title: Long-term Effectiveness and Safety of Empagliflozin-based Quadruple Oral Antidiabetic Agents Therapy Compared to Basal Insulin-based Combination Therapy in Patients With Type 2 Diabetes
Brief Title: Empagliflozin-based Quadruple Therapy vs Basal Insulin-based Therapy
Acronym: LUCID
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chungbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Eu Jeong Ku, Clinical Associate Professor, Chungbuk National University Hospital
Other Study IDs: CBNUH-LUCID
Record Dates: First submitted 2021-11-01; First posted 2021-11-02 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes mellitus; Sodium-glucose co-transporter 2 inhibitor; Empagliflozin; Insulin glargine; Insulin degludec
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Triple OADs failure: Inadequatelly controlled type 2 diabetes patients despite triple combination therapy with metformin, glimepiride, and DPP-4 inhibitor
  Interventions: Drug: Empagliflozin 25 MG; Drug: INS

INTERVENTIONS:
Drug: Empagliflozin 25 MG — Empagliflozin 25mg/day add-on to triple combination oral antidiabetic agents consisted with metformin, glimepiride, and DPP4 inhibitor
Drug: INS — Basal insulin add on the background OADs
  Other Names: Basal insulin

SUMMARY:
This study aimed to evaluate the long-term effectiveness and safety of the empagliflozin as add-on thearpy compared to basal insulin-based antidiabetic agents (OADs) combination therapy in patients with type 2 diabetes inadequately controlled on triple OADs in a real clinical practice.

DETAILED DESCRIPTION:
This study aimed to evaluate the long-term effectiveness and safety of the empagliflozin as add-on thearpy compared to basal insulin-based antidiabetic agents (OADs) combination therapy in patients with type 2 diabetes inadequately controlled on triple OADs in a real clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Inadequately controlled with triple OADs (metformin, glimepiride, dipeptidyl peptidase-4 inhibitor) showing HbA1c 7.5-12.0%

Exclusion Criteria:

* Type 1 diabetes
* Gestional diabetes
* Diabetes due to secondary causes
* Receiving anticancer treatment
* Receiving glucocorticoids or immune-suppressants
* Have been treated with sodium glucose co-transporter 2 inhibitors for more than 7 consecutive days within 3 months before entering the study
* Have been treated with any type of insulin for more than 7 consecutive days within 3 months before entering the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetes, uncontrolled with triple OADs
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Changes in HbA1c From Baseline to months 36 | Baseline, month 36 (3-year)
  Changes in HbA1c From Baseline to months 36 (3-year)

SECONDARY OUTCOMES:
Achievement of target HbA1c | Baseline, month 36
  Percentage of Patients Who Achieved Glycemic Target of HbA1c at month 36
Changes in HbA1c | Baseline, month 3, 6, 12, 18, 24, 30
  Changes in HbA1c From Baseline to each time frame
Changes in FPG | Baseline, month 3, 6, 12, 18, 24, 30, 36
  Changes in fasting plasma glucose level from baseline to each month
Changes in lipid profiles | Baseline, month 36
  Changes in total cholesterol, triglyceride, HDL-cholesterol and LDL cholesterol from baseline to month 36
Changes in body weight | Baseline, month 36
  Changes in body weight from baseline to month 36
Changes in blood pressure | Baseline, month 36
  Changes in systolic and diastolic blood pressure from baseline to month 36
Percentage of patients with hypoglycemic episodes | Baseline, month 36
  All episodes consistent with hypoglycemia with or without a confirmatory blood glucose reading were collected.
Percentage of patients with at least 1 episode of genitourinary tract infections | Baseline, month 36
  Percentage of Patients With At Least 1 Episode of Genitourinary Tract Infections

CONTACTS AND LOCATIONS:
Overall Officials: Eu Jeong Ku, MD, PhD, Principal Investigator — Chungbuk National University Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ku EJ, Oh TK. Long-Term Effectiveness of Quadruple Combination Therapy with Empagliflozin Versus Basal Long-Acting Insulin Therapy in Patients with Type 2 Diabetes: 3-Year Retrospective Observational Study. Diabetes Ther. 2023 Sep;14(9):1471-1479. doi: 10.1007/s13300-023-01437-x. Epub 2023 Jun 27. PMID 37369826